CLINICAL TRIAL: NCT04152005
Title: Analysis of Endothelin Concentrations in a Population With Cardiovascular Disease and Periodontitis
Brief Title: Endothelin Concentrations in a Population With Cardiovascular Disease and Periodonitis
Status: Completed | Type: Observational
Sponsor: University of Messina (Other)
Responsible Party: Principal Investigator, Gaetano Isola, DDS, PhD, Assistant Professor, University of Messina
Other Study IDs: 10-918-10
Record Dates: First submitted 2019-11-01; First posted 2019-11-05 (Actual); Last update posted 2019-11-06 (Actual); Status verified 2019-11

CONDITIONS: Serum; Disease
MeSH Terms: conditions — Disease | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Control: Evaluation of ET-1 level and correlation of ET-1 levels with periodontal and cardiovascular disease
  Interventions: Other: Observation
- Periodontitis: Evaluation of ET-1 level and correlation of ET-1 levels with periodontal and cardiovascular disease
  Interventions: Other: Observation
- Cardiovascular: Evaluation of ET-1 level and correlation of ET-1 levels with periodontal and cardiovascular disease
  Interventions: Other: Observation
- Periodontitis+Cardiovascular: Evaluation of ET-1 level and correlation of ET-1 levels with periodontal and cardiovascular disease
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Evaluation of ET-1 level and correlation of ET-1 levels with periodontal and cardiovascular disease

SUMMARY:
Recently, a key role played in the ethiology of periodontitis has been highlighted by a Endothelin (ET-1). ET1 possess the ability to express surface antigens of endothelial and hematopoietic stem cells and to assist in maintaining vascular integrity and the repair mechanism of the endothelium. ET originate from bone marrow

DETAILED DESCRIPTION:
The aim of the present study was to investigate the association between ET-1 in patients with periodontitis. Furthermore, the objective was to determine if the periodontal status influenced ET-1 levels.

ELIGIBILITY:
Inclusion Criteria:

* Presence of at least 16 teeth
* CP with a minimum of 40% of sites with a clinical attachment level (CAL)

  ≥2mm and probing depth (PD) ≥4mm;
* Presence of at least ≥2 mm of crestal alveolar bone loss verified on digital periapical radiographs
* Presence of ≥40% sites with bleeding on probing (BOP)

Exclusion Criteria:

* Intake of contraceptives
* Intake of immunosuppressive or anti-inflammatory drugs throughout the last three months prior to the study
* Status of pregnancy or lactation
* Previous history of excessive drinking
* Allergy to local anaesthetic
* Intake of drugs that may potentially determine gingival hyperplasia such as Hydantoin, Nifedipine, Cyclosporin A or similar drugs.

Ages: 21 Years to 71 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 34 patients with CP, 34 patients with CHD, 34 patients with CP+CHD, and 34 healthy subjects were finally enrolled
Sampling Method: Non-Probability Sample
Enrollment: 165 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-09-25 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Evaluation of ET-1 levels | 1 year
  Correlation of ET-1 levels with periodontal and cardiovascular disease

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Matarese, Study Director — University of Messina
Locations (1):
- University of Messina, Messina, Italy

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD, all IPD that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: 5 years
Access Criteria: IRB university of messina